CLINICAL TRIAL: NCT02783274
Title: Actis Total Hip System 2 Year Follow-up
Acronym: Actis14014
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14014
Record Dates: First submitted 2016-05-23; First posted 2016-05-26 (Estimated); Results first posted 2025-05-22 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis; Traumatic Arthritis; Rheumatoid Arthritis; Congenital Hip Dysplasia; Avascular Necrosis of the Femoral Head; Acute Traumatic Fracture of the Femoral Head or Neck; Certain Cases of Ankylosis; Non-union of Femoral Neck Fractures; Certain High Sub-Capital & Femoral Neck Fractures in Elderly
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Hip Dislocation, Congenital; Femur Head Necrosis

STUDY DESIGN:
Intervention Model Description: Single cohort of Total Hips and the protocol also includes a single cohort for Hemi-hips. No comparisons are made to comparator devices, no randomization (open label). gathering data for a Post-market clinical follow-up study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Actis Total Hip System (Other): The Actis DuoFix Femoral Stem can be used for both a Total and Hemi-hip Replacement
  Interventions: Device: Actis Total Hip System

INTERVENTIONS:
Device: Actis Total Hip System — Total Hip Replacement and Hemi-hip Replacement
  Other Names: Actis DuoFix Femoral Stem

SUMMARY:
Two-year (2 year) information regarding the performance of the commercially available Actis™ Total Hip System in order to obtain and evaluate the clinical outcomes on a series of cementless primary total hip arthroplasty (THA) and hemi-hip arthroplasty procedures using clinical, radiographic and device and procedure related adverse event assessments.

DETAILED DESCRIPTION:
A minimum of 10 study sites.

A prospective, uncontrolled, non-randomized, multicenter study.

A total of 255 Subjects to include a minimum of 225 Primary THA Subjects and a Sub-group with a minimum of 30 hemi-hip arthroplasty Subjects will be prospectively enrolled into the study. All Subjects will be seen for a preoperative clinic visit at the time of consent, and evaluated at the time of surgery, 6 weeks (28-70 days), 3 months (71-132 days), minimum 1 year (304-668 days), and minimum 2 years (669-1,763 days) postoperatively.

ELIGIBILITY:
Inclusion Criteria:

Total primary hip replacement is indicated in the following conditions:

1. A severely painful and/or disable joint from osteoarthritis, traumatic arthritis, rheumatoid arthritis, or congenital hip dysplasia.
2. Avascular necrosis of the femoral head.
3. Acute traumatic fracture of the femoral head or neck.
4. Certain cases of ankylosis.

   Hemi-hip arthroplasty is indicated in the following conditions:
5. Acute fracture of the femoral head or neck that cannot be appropriately reduced and treated with internal fixation.
6. Fracture dislocation of the hip that cannot be appropriately reduced and treated with internal fixation.
7. Avascular necrosis of the femoral head.
8. Non-union of femoral neck fractures.
9. Certain high sub-capital and femoral neck fractures in the elderly.
10. Degenerative arthritis involving only the femoral head in which the acetabulum does not require replacement.
11. Pathology involving only the femoral head in which the acetabulum does not require replacement.

    Further inclusion criteria for individuals who, in the opinion of the Principal Investigator, are suitable candidates for using the devices specified in this protocol and they are as follows:
12. Individuals who are able to speak, read, and comprehend the informed patient consent (IPC) document and willing and able to provide informed patient consent for participation in the study and have authorized the transfer of his/her information to DePuy Synthes (Joint Reconstruction).
13. Individuals who are willing and able to return for follow-up as specified by the study protocol.
14. Individuals who are a minimum age of 21 years at the time of consent.
15. Individuals who are not bedridden.
16. Individuals who are willing and able to complete the Subject Hip Outcomes questionnaires (i.e., FJS-12, HOOS and Hip Evaluation) as specified by the study protocol.
17. Individuals interested in participating in the parallel and optional Patient Activity Tracking portion of the study are required to link the Patient Activity Tracking device to their own well-functioning smartphone (i.e., iPhone or Android phone) via a downloaded mobile application (i.e., ActiTrak™). If a Subject does not have a smartphone, and would like to participate in the Patient Activity Tracking portion of the study, the Sponsor will be able to provide an Android type tablet to which the required app can be downloaded.
18. Individuals interested in participating in the optional Patient Activity Tracking (ActiTrak™) portion of the study must be willing to wear the Patient Activity Tracking device from the time of consent preoperative (if possible, based on date of consent) and for 3 months postoperative.
19. Individuals interested in participating in the optional Patient Activity Tracking (ActiTrak™) portion of the study must have the ability to return at the 3 month follow-up visit in order to return the Patient Activity Tracking device, and if applicable, the Sponsor's Android tablet back to the study site.

Exclusion Criteria:

* Subjects will be excluded if in the opinion of the Investigator, the individual meets any of the following exclusions:

  1. Active local or systemic infection.
  2. Loss of musculature, neuromuscular compromise or vascular
  3. Poor bone quality, such as osteoporosis, where in the surgeon's opinion, there could be considerable migration of the prosthesis or a significant chance of fracture of the femoral shaft and/or the lack of adequate bone to support the implant(s).
  4. Charcot's or Paget's disease.
  5. For hemi-hip arthroplasty, any pathological condition of the acetabulum, such as distorted acetabuli with irregularities, protrusion acetabuli (arthrokatadysis), or migrating acetabuli, that would preclude the use of the natural acetabulum as an appropriate articular surface for the hemi-hip prosthesis.
  6. The Subject is a woman who is pregnant or lactating.
  7. Existing contralateral hip that was implanted less than 6 months from the date of surgery at the time of consent into this study.
  8. Subjects requiring a simultaneous bilateral hip at the time of consent will be excluded; there can be only one Actis™ study hip. This also means that even if another hip system is used for the contralateral hip during simultaneous THAs, the Subject will be excluded. As noted above, Subjects who have an existing contralateral total hip replacement greater than 6 months postoperatively at the time of consent may be entered into this study if they qualify based upon the eligibility criteria and the approved labeling requirements.
  9. Subject had a contralateral amputation.
  10. Subject has participated in a clinical investigation with an investigational product (drug or device) in the last three months.
  11. Subject is currently involved in any personal injury litigation, medical-legal or worker's compensation claims.
  12. Subject, in the opinion of the Investigator, is a drug or alcohol abuser or has a psychological disorder that could affect their ability to complete patient reported questionnaires or be compliant with follow-up requirements.
  13. Subject was diagnosed and is taking prescription medications to treat a muscular disorder that limits mobility due to severe stiffness and pain such as fibromyalgia or polymyalgia.
  14. Subject has a medical condition with less than 2 years of life expectancy. Note: Diabetes, at present, has not been established as a contraindication. However, because of the increased risk for complications such as infection, slow wound healing, etc., the physician should carefully consider the advisability of hip replacement in the severely diabetic patient.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah German, BS, Study Director — DePuy Synthes
Locations (9):
- United States (9):
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Rochester, Minnesota
  - Lebanon, New Hampshire
  - New York, New York
  - Charlotte, North Carolina
  - Philadelphia, Pennsylvania
  - Austin, Texas
  - Renton, Washington

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: https://yoda.yale.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All eligible patients were asked if they were interested in study participation. 266 Hips in 266 Patients were enrolled into the study.
Units Other Than Participants: Hips
Period: Overall Study
Arm/Group | Actis Total Hip System
Started | 266; 266 Hips
Treated | 255; 255 Hips
Total Hip Replacement Participants (THA) | 232; 232 Hips
Hemi-hip Replacement Participants (HHA) | 23; 23 Hips
Completed | 191; 191 Hips
Not Completed | 75; 75 Hips
Not completed — Withdrawal by Subject | 16
Not completed — Physician Decision | 6
Not completed — Death | 9
Not completed — Lost to Follow-up | 22
Not completed — Other | 22

BASELINE CHARACTERISTICS:
Population: All Implanted Participants (n=255)
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 255
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age in years of implanted participants (n=255) Population: All implanted participants (n=255)
  Years | 62.6 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender of implanted participants (n=255) Population: Implanted Participants
  Participants
    Female | 119
    Male | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity of implanted participants Population: Implanted Participants
  Participants
    Hispanic or Latino | 8
    Not Hispanic or Latino | 247
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of implanted Participants Population: Implanted Participants
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 1
    Black or African American | 20
    White | 231
    More than one race | 2
    Unknown or Not Reported | 1
Implanted Participant Primary Diagnosis [Count of Participants; unit: Participants] — Primary Diagnosis of Implanted Participants Population: Implanted Participants
  Participants
    Acute Fracture | 22
    Avascular Necrosis | 8
    Degenerative Joint Disease | 41
    Hip Dysplasia | 2
    Osteoarthritis | 179
    Rheumatoid Arthritis | 1
    Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Harris Hip Score- THA Subjects Per Protocol at 2 Years
Description: The Harris Hip Score (HHS) is a standardized tool used to evaluate hip pain, function, and mobility. The HHS is score from 0 to 100, with higher scores indicating better outcomes. A score of less than 70 is considered poor, 70-80 is fair, 80-90 is good, 90-100 is excellent.
Time Frame: 2 Years
Population: All implanted participants who attended their 2-year clinical evaluation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 166
units on a scale | 95.7 (9.3)

2. Primary Outcome: Harris Hip Score- HHA Subjects Per Protocol at 2 Years
Description: as for outcome 1
Time Frame: 2 Years
Population: All implanted participants who attended their 2-year clinical evaluation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 5
units on a scale | 83.2 (15.3)

3. Secondary Outcome: Harris Hip Score- THA Subjects Per Protocol at 3 Months
Description: as for outcome 1
Time Frame: 3 months
Population: All implanted participants who attended their 3-month clinical evaluation
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 189
Units on a scale | 93.5 (8.7)

4. Secondary Outcome: Harris Hip Score- HHA Subjects Per Protocol at 3 Months
Description: as for outcome 1
Time Frame: 3 months
Population: All implanted participants who attended their 3-month clinical evaluation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 9
units on a scale | 85.3 (14.3)

5. Secondary Outcome: Harris Hip Score- THA Subjects Per Protocol at 1 Year
Description: as for outcome 1
Time Frame: 1 Year
Population: All implanted participants who attended their 1-year clinical evaluation
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 186
Units on a scale | 95.7 (9.0)

6. Secondary Outcome: Harris Hip Score- HHA Subjects Per Protocol at 1 Year
Description: as for outcome 1
Time Frame: 1 Year
Population: All implanted participants who attended their 1-year clinical evaluation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 5
units on a scale | 85.8 (12.6)

7. Secondary Outcome: Post-Operative 2-Year Device Survivorship- THA Subjects Safety Population
Description: Device survivorship at 2 years post-operatively is a secondary endpoint in this study. A revision is defined as a revision for any reason and device survival is defined as the lack of revision. A 2-year Kaplan-Meier survivorship estimate of the Actis Hip System in implanted hips is provided.
Time Frame: 2 Years
Population: All THA implanted Participants
Measure: Number (95% Confidence Interval); unit: Percentage of hip Implants
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 255
Number analyzed (Hips) | 255
Percentage of hip Implants | 97.7 [94.5 to 99.0]

8. Secondary Outcome: Post-Operative 2-Year Femoral Stem Survivorship- THA Subjects Safety Population
Description: A stem revision is defined as any stem revision for any reason and device survival is defined as the lack of revision. A 2-year Kaplan-Meier survivorship estimate of the Actis Hip System in implanted hips is provided.
Time Frame: 2 Years
Population: All THA Implanted Participants
Measure: Number (95% Confidence Interval); unit: Percentage of hip Implants
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 255
Number analyzed (Hips) | 255
Percentage of hip Implants | 99.6 [96.9 to 99.9]

9. Secondary Outcome: Acetabular Shell Version at 2-years Postoperatively- THA Subjects Per Protocol
Description: Acetabular cup version is the angle formed between the axis of the implant and the coronal plane of the body. Acetabular version typically ranges between 11.5 and 28.5 degrees.
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 166
Number analyzed (Hips) | 166
Degrees | 25.9 (3.89)

10. Secondary Outcome: Acetabular Shell Inclination at 2-years Postoperatively- THA Subjects Per Protocol
Description: Acetabular cup inclination is the angle between the longitudinal axis of the patient and a perpendicular line to the major axis of the cup projection. The target acetabular cup inclination is between 30-50 degrees
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 168
Number analyzed (Hips) | 16
Degrees | 39.9 (4.87)

11. Secondary Outcome: Number of Participants With >4 Degrees Change in Acetabular Cup Inclination Angle at 2 Years Postoperatively - THA Subjects
Description: Number of participants with greater than (>) 4 degrees change in acetabular cup inclination angle at 2 years postoperatively was reported.
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 168
Participants | 1 [lower limit 4.87]

12. Secondary Outcome: Number of Participants With Acetabular Shell Migration >2mm at 2 Years Postoperatively - THA Subjects Per Protocol
Description: Number of participants with acetabular shell migration >2mm at 2 years postoperatively were reported. Acetabular migration is the superior migration of the implant within the pelvic bone.
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 168
Participants | 0 [lower limit 4.87]

13. Secondary Outcome: Acetabular Radiolucent Lines- THA Subjects Per Protocol
Description: Radiolucent lines are seen on x-rays and represent an area that is absent of bone. Radiolucent lines seen adjacent to an implant may suggest a lack on bone ingrowth or possible loosening of the implant. Radiolucent lines greater than 1mm wide were considered reportable for this study.
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 168
Number analyzed (Hips) | 168
Hips | 5 [lower limit 4.87]

14. Secondary Outcome: Acetabular Osteolysis- THA Subjects Per Protocol
Description: Osteolysis is seen on x-rays and represent an area where bone has been resorbed by the body in response to small particles of debris that are created as an implant wears over time. Osteolysis greater than 5mm was considered to be reportable for this study.
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 168
Number analyzed (Hips) | 168
Hips | 0 [lower limit 4.87]

15. Secondary Outcome: Acetabular Sclerotic Lines- THA Subjects Per Protocol
Description: Acetabular sclerotic lines are seen on x-rays and are radio-dense areas of bone that have remodeled due to loads close to the implant.
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 168
Number analyzed (Hips) | 168
Hips | 38 [lower limit 4.87]

16. Secondary Outcome: Acetabular Porous Coating Integrity- THA Subjects Per Protocol
Description: Acetabular Cup Porous Coating Integrity is defined as the presence of one or more beads of the porous coating observed away from the component in the soft tissue adjacent to the device.
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 168
Number analyzed (Hips) | 168
Hips | 0 [lower limit 4.87]

17. Secondary Outcome: Femoral Stem Position- THA Subjects Per Protocol
Description: Femoral stem position is categorized as neutral, valgus, or varus. A neutral stem is centered within the femoral canal that runs through the center of the femur's long axis. A valgus femoral stem is positioned slightly towards the medial side of the femoral canal, and a varus femoral stem is positioned slightly towards the lateral side of the femoral canal.
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 168
Number analyzed (Hips) | 168
Hips
  Neutral | 160 [lower limit 4.87]
  Valgus | 3 [lower limit 4.87]
  Varus | 5 [lower limit 4.87]

18. Secondary Outcome: Femoral Stem Position- HHA Subjects Per Protocol
Description: as for outcome 17
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 6
Number analyzed (Hips) | 6
Hips
  Neutral | 5 [lower limit 4.87]
  Valgus | 0 [lower limit 4.87]
  Varus | 1 [lower limit 4.87]

19. Secondary Outcome: Number of Participants With Femoral Stem Tilt - THA Subjects Per Protocol
Description: Number of participants with femoral stem tilt were reported. Femoral stem tilt is a measurement taken at each post-operative year and compared against baseline images collected at 6-weeks post-operative. The measurement captures changes in the position of the femoral stem over time.
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 168
Participants | 1

20. Secondary Outcome: Number of Participants With Femoral Stem Tilt- HHA Subjects Per Protocol
Description: as for outcome 19
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 6
Participants | 0

21. Secondary Outcome: Number of Participants With Femoral Stem Subsidence- THA Subjects Per Protocol
Description: Femoral stem subsidence is the inferior movement of the stem within the femoral canal. Subsidence greater than 2 mm was considered reportable for this study.
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 168
Participants | 0

22. Secondary Outcome: Number of Participants With Femoral Stem Subsidence- HHA Subjects Per Protocol
Description: as for outcome 21
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 6
Participants | 0

23. Secondary Outcome: Femoral Stem Heterotopic Ossification- THA Subjects Per Protocol
Description: Heterotopic ossification is the abnormal formation of bone in soft tissues, such as muscles, tendons, or ligaments and can occur around the hip joint, leading to pain, stiffness, and restricted range of motion. It is grade as Class 0 through Class IV, with Class 0 being least impactful and Class IV being most impactful.
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 168
Number analyzed (Hips) | 168
Hips
  Class 0 | 98
  Class I | 55
  Class II | 11
  Class III | 3
  Unable to Assess | 1

24. Secondary Outcome: Femoral Stem Heterotopic Ossification- HHA Subjects Per Protocol
Description: as for outcome 23
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 6
Number analyzed (Hips) | 6
Hips
  Class 0 | 2
  Class I | 2
  Class II | 0
  Class III | 2

25. Secondary Outcome: Femoral Radiolucent Lines- THA Subjects Per Protocol
Description: Radiolucencies are seen on x-rays and represent an area that is absent of bone. Radiolucent lines seen adjacent to an implant may suggest a lack of bone ingrowth into the implant or possible loosening of the implant.
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 168
Number analyzed (Hips) | 168
Hips | 1

26. Secondary Outcome: Femoral Radiolucent Lines- HHA Subjects Per Protocol
Description: as for outcome 25
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 6
Number analyzed (Hips) | 6
Hips | 0

27. Secondary Outcome: Femoral Osteolysis- THA Subjects Per Protocol
Description: as for outcome 14
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 168
Number analyzed (Hips) | 168
Hips | 0

28. Secondary Outcome: Femoral Osteolysis- HHA Subjects Per Protocol
Description: as for outcome 14
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 6
Number analyzed (Hips) | 6
Hips | 0

29. Secondary Outcome: Femoral Stem Sclerotic Lines- THA Subjects Per Protocol
Description: Sclerotic lines are seen on x-rays and are radio-dense areas of bone that have remodeled due to loads close to the implant.
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 168
Number analyzed (Hips) | 168
Hips | 102

30. Secondary Outcome: Femoral Stem Sclerotic Lines- HHA Subjects Per Protocol
Description: as for outcome 29
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 6
Number analyzed (Hips) | 6
Hips | 5

31. Secondary Outcome: Femoral Stem Porous Coating Integrity- THA Subjects Per Protocol
Description: as for outcome 16
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 168
Number analyzed (Hips) | 168
Hips | 0

32. Secondary Outcome: Femoral Stem Porous Coating Integrity- HHA Subjects Per Protocol
Description: Femoral Stem Porous Coating Integrity is defined as the presence of one or more beads of the porous coating observed away from the component in the soft tissue adjacent to the device.
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 6
Number analyzed (Hips) | 6
Hips | 0

33. Secondary Outcome: Femoral Stem Calcar Resorption- THA Subjects Per Protocol
Description: Femoral calcar resorption occurs when the bone around the prosthesis is partially shielded from bearing loads and begins to resorb
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 168
Number analyzed (Hips) | 168
Hips | 73

34. Secondary Outcome: Femoral Stem Calcar Resorption- HHA Subjects Per Protocol
Description: as for outcome 33
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 6
Number analyzed (Hips) | 6
Hips | 3

35. Secondary Outcome: Femoral Stem Calcar Fracture- THA Subjects Per Protocol
Description: Near the top of the femur is a region of bone called the calcar femorale that provides strength to the femur when compressive forces are applied. During preparation of the femur to receive the femoral implant there is the possibility of fractures occurring in this region.
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 168
Number analyzed (Hips) | 168
Hips | 3

36. Secondary Outcome: Femoral Stem Calcar Fracture- HHA Subjects Per Protocol
Description: as for outcome 35
Time Frame: 2 Years
Population: All implanted participants with radiographs on file at the 2-year study visit
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 6
Number analyzed (Hips) | 6
Hips | 0

37. Secondary Outcome: Perceived Leg Length Discrepancy- THA Subjects Per Protocol
Description: The number of subjects who perceived a Leg Length Discrepancy at Two Years
Time Frame: 2 Years
Population: Implanted subjects who attended the 2-year clinic visit and answered this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 163
Participants | 11

38. Secondary Outcome: Perceived Leg Length Discrepancy- HHA Subjects Per Protocol
Description: The number of subjects who perceived a Leg Length Discrepancy at Two Years
Time Frame: 2 Years
Population: Implanted subjects who attended the 2-year clinic visit and answered this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 2
Participants | 0

39. Secondary Outcome: Number of Participants With True Leg Length Discrepancy- THA Subjects Per Protocol
Description: True LLD is defined as a difference of 3 cm or greater as reviewed via postoperative radiographs. The measurement is the distance between the superior-most aspects of the left and right femoral heads
Time Frame: 2 Years
Population: Implanted subjects with a 2-year radiograph on file
Measure: Count of Participants; unit: Participants
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 163
Participants | 0

40. Secondary Outcome: Number of Participants With True Leg Length Discrepancy- HHA Subjects Per Protocol
Description: as for outcome 39
Time Frame: 2 Years
Population: Implanted subjects with a 2-year radiograph on file
Measure: Count of Participants; unit: Participants
Arm/Group | Actis Total Hip System
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the course of the study and continued until the 2-year interval when the study closed
Description: Adverse events were collected throughout the course of the study and continued until the 2-year interval when the study closed
Arm/Group | Actis Total Hip System
All-Cause Mortality (participants affected / at risk) | 9/255
Serious Adverse Events (participants affected / at risk) | 8/255
Other Adverse Events (participants affected / at risk) | 22/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Actis Total Hip System (N=255)
Wound Abscess (Infections and infestations) | 1 (2)
Post procedural infection (Infections and infestations) | 2 (2)
Wound decomposition (Injury, poisoning and procedural complications) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Medical device site joint infection (Infections and infestations) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Device dislocation (Product Issues) | 1 (1)
Device failure (Product Issues) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Actis Total Hip System (N=255)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (12)
Joint dislocation (Injury, poisoning and procedural complications) | 5 (7)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Impaired healing (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT02783274/Prot_SAP_000.pdf